CLINICAL TRIAL: NCT04811573
Title: Bioequivalence of Three Different Tablet Formulations of 30 mg of Apremilast (EU-sourced Otezla® vs. US-sourced Otezla® vs. Japan-sourced Otezla®) Administered in Healthy Male and Female Subjects in the Fasted State as Well as (for EU-sourced Otezla® vs. US-sourced Otezla®) in the Fed State (an Open-label, Randomised, Single-dose, Five-period, Ten-sequence Crossover Study)
Brief Title: A Study in Healthy People to Compare 3 Different Formulations of Apremilast Tablets Taken With or Without Food
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: due to company decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1407-0041; 2019-005037-37 (EudraCT Number)
Record Dates: First submitted 2021-03-22; First posted 2021-03-23 (Actual); Results first posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2022-08

CONDITIONS: Healthy
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Intervention Model Description: Five-period, ten-sequence crossover trial.
  Periods:
  (A): EU-sourced Otezla - fasted condition (B): US-sourced Otezla - fasted condition (C): EU-sourced Otezla - fed condition (C): US-sourced Otezla - fed condition (E): Japan-sourced Otezla - fasted condition
  Sequences: see Arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (10):
- EU-Otezla fasted(A)/ Japan-Otezla fasted(E)/ US-Otezla fasted(B)/ US-Otezla fed(D)/ EU-Otezla fed(C) (Experimental): Treatment sequence AEBDC is applied. The 5 treatments were separated by a washout period of at least 5 days.
  Interventions: Drug: EU-sourced Otezla®; Drug: US-sourced Otezla®; Drug: Japan-sourced Otezla®
- US-Otezla fasted(B)/ EU-Otezla fasted(A)/ EU-Otezla fed(C)/ Japan-Otezla fasted(E)/ US-Otezla fed(D) (Experimental): Treatment sequence BACED is applied. The 5 treatments were separated by a washout period of at least 5 days.
  Interventions: Drug: EU-sourced Otezla®; Drug: US-sourced Otezla®; Drug: Japan-sourced Otezla®
- EU-Otezla fed(C)/US-Otezla fasted(B)/US-Otezla fasted(D)/EU-Otezla fasted(A)/ Japan-Otezla fasted(E) (Experimental): Treatment sequence CBDAE is applied. The 5 treatments were separated by a washout period of at least 5 days.
  Interventions: Drug: EU-sourced Otezla®; Drug: US-sourced Otezla®; Drug: Japan-sourced Otezla®
- US-Otezla fed(D)/ EU-Otezla fed(C)/ Japan-Otezla fasted(E)/ US-Otezla fasted(B)/ EU-Otezla fasted(A) (Experimental): Treatment sequence DCEAB is applied. The 5 treatments were separated by a washout period of at least 5 days.
  Interventions: Drug: EU-sourced Otezla®; Drug: US-sourced Otezla®; Drug: Japan-sourced Otezla®
- Japan-Otezla fasted(E)/ US-Otezla fed(D)/ EU-Otezla fasted(A)/EU-Otezla fed(C)/ US-Otezla fasted(B) (Experimental): Treatment sequence EDACB is applied. The 5 treatments were separated by a washout period of at least 5 days.
  Interventions: Drug: EU-sourced Otezla®; Drug: US-sourced Otezla®; Drug: Japan-sourced Otezla®
- EU-Otezla fasted(A)/ US-Otezla fasted(B)/ Japan-Otezla fasted(E)/ EU-Otezla fed(C)/ US-Otezla fed(D) (Experimental): Treatment sequence ABECD is applied. The 5 treatments were separated by a washout period of at least 5 days.
  Interventions: Drug: EU-sourced Otezla®; Drug: US-sourced Otezla®; Drug: Japan-sourced Otezla®
- US-Otezla fasted(B)/ EU-Otezla fed(C)/ EU-Otezla fasted(A)/ US-Otezla fed(D)/ Japan-Otezla fasted(E) (Experimental): Treatment sequence BCADE is applied. The 5 treatments were separated by a washout period of at least 5 days.
  Interventions: Drug: EU-sourced Otezla®; Drug: US-sourced Otezla®; Drug: Japan-sourced Otezla®
- EU-Otezla fed(C)/ US-Otezla fed(D)/ US-Otezla fasted(B)/ Japan-Otezla fasted(E)/ EU-Otezla fasted(A) (Experimental): Treatment sequence CDBEA is applied. The 5 treatments were separated by a washout period of at least 5 days.
  Interventions: Drug: EU-sourced Otezla®; Drug: US-sourced Otezla®; Drug: Japan-sourced Otezla®
- US-Otezla fed(D)/ Japan-Otezla fasted(E)/ EU-Otezla fed(C)/ EU-Otezla fasted(A)/ US-Otezla fasted(B) (Experimental): Treatment sequence DECAB is applied. The 5 treatments were separated by a washout period of at least 5 days.
  Interventions: Drug: EU-sourced Otezla®; Drug: US-sourced Otezla®; Drug: Japan-sourced Otezla®
- Japan-Otezla fasted(E)/ EU-Otezla fasted(A)/ US-Otezla fed(D)/ US-Otezla fasted(B)/ EU-Otezla fed(C) (Experimental): Treatment sequence EADBC is applied. The 5 treatments were separated by a washout period of at least 5 days.
  Interventions: Drug: EU-sourced Otezla®; Drug: US-sourced Otezla®; Drug: Japan-sourced Otezla®

INTERVENTIONS:
Drug: EU-sourced Otezla® — Test product
  Other Names: Apremilast
Drug: US-sourced Otezla® — Reference product 1
  Other Names: Apremilast
Drug: Japan-sourced Otezla® — Reference product 2
  Other Names: Apremilast

SUMMARY:
The aim of this trial is to establish bioequivalence between EU-, US- and Japan-sourced Otezla® tablet formulations to assure comparability of results from Phase III trials of BI 730357 (new oral agent for treatment of psoriasis as well as other T helper 17 cells (Th17)-mediated diseases) regardless of whether only the EU-sourced Otezla® or EU and US-sourced Otezla®/Japan-sourced Otezla® have been used as an active comparator.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects, or female subjects who meet any of the following criteria for a highly effective contraception from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal), plus condom
  * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom
  * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy or bilateral occlusion)
  * Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of Follicle-stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label, randomised, single-dose, five-period, ten-sequence crossover study was to compare the test treatment (EU-sourced Otezla) to the reference treatments US-sourced Otezla and Japan-sourced Otezla) under fasting and fed conditions.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- EU-Otezla Fasted(A)/ Japan-Otezla Fasted(E)/ US-Otezla Fasted(B)/ US-Otezla Fed(D)/ EU-Otezla Fed(C): Treatment sequence AEBDC was applied:
  EU-Otezla fasted(A): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  US-Otezla fasted(B): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  EU-Otezla fed(C): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  US-Otezla fed(D): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  Japan-Otezla fasted(E): One Japan-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  The 5 treatments were separated by a washout period of at least 5 days.
- US-Otezla Fasted(B)/ EU-Otezla Fasted(A)/ EU-Otezla Fed(C)/ Japan-Otezla Fasted(E)/ US-Otezla Fed(D): Treatment sequence BACED was applied with the following treatments:
  EU-Otezla fasted(A): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  US-Otezla fasted(B): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  EU-Otezla fed(C): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  US-Otezla fed(D): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  Japan-Otezla fasted(E): One Japan-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  The 5 treatments were separated by a washout period of at least 5 days.
- EU-Otezla Fed(C)/US-Otezla Fasted(B)/US-Otezla Fed(D)/EU-Otezla Fasted(A)/ Japan-Otezla Fasted(E): Treatment sequence CBDAE was applied with the following treatments:
  EU-Otezla fasted(A): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  US-Otezla fasted(B): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  EU-Otezla fed(C): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  US-Otezla fed(D): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  Japan-Otezla fasted(E): One Japan-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  The 5 treatments were separated by a washout period of at least 5 days.
- US-Otezla Fed(D)/ EU-Otezla Fed(C)/ Japan-Otezla Fasted(E)/ US-Otezla Fasted(B)/ EU-Otezla Fasted(A): Treatment sequence DCEAB was applied with the following treatments:
  EU-Otezla fasted(A): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  US-Otezla fasted(B): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  EU-Otezla fed(C): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  US-Otezla fed(D): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  Japan-Otezla fasted(E): One Japan-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  The 5 treatments were separated by a washout period of at least 5 days.
- Japan-Otezla Fasted(E)/ US-Otezla Fed(D)/ EU-Otezla Fasted(A)/EU-Otezla Fed(C)/ US-Otezla Fasted(B): Treatment sequence EDACB was applied with the following treatments:
  EU-Otezla fasted(A): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  US-Otezla fasted(B): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  EU-Otezla fed(C): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  US-Otezla fed(D): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  Japan-Otezla fasted(E): One Japan-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  The 5 treatments were separated by a washout period of at least 5 days.
- EU-Otezla Fasted(A)/ US-Otezla Fasted(B)/ Japan-Otezla Fasted(E)/ EU-Otezla Fed(C)/ US-Otezla Fed(D): Treatment sequence ABECD was applied with the following treatments:
  EU-Otezla fasted(A): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  US-Otezla fasted(B): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  EU-Otezla fed(C): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  US-Otezla fed(D): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  Japan-Otezla fasted(E): One Japan-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  The 5 treatments were separated by a washout period of at least 5 days.
- US-Otezla Fasted(B)/ EU-Otezla Fed(C)/ EU-Otezla Fasted(A)/ US-Otezla Fed(D)/ Japan-Otezla Fasted(E): Treatment sequence BCADE was applied with the following treatments:
  EU-Otezla fasted(A): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  US-Otezla fasted(B): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  EU-Otezla fed(C): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  US-Otezla fed(D): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  Japan-Otezla fasted(E): One Japan-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  The 5 treatments were separated by a washout period of at least 5 days.
- EU-Otezla Fed(C)/ US-Otezla Fed(D)/ US-Otezla Fasted(B)/ Japan-Otezla Fasted(E)/ EU-Otezla Fasted(A): Treatment sequence CDBEA was applied with the following treatments:
  EU-Otezla fasted(A): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  US-Otezla fasted(B): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  EU-Otezla fed(C): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  US-Otezla fed(D): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  Japan-Otezla fasted(E): One Japan-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  The 5 treatments were separated by a washout period of at least 5 days.
- US-Otezla Fed(D)/ Japan-Otezla Fasted(E)/ EU-Otezla Fed(C)/ EU-Otezla Fasted(A)/ US-Otezla Fasted(B): Treatment sequence DECAB was applied with the following treatments:
  EU-Otezla fasted(A): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  US-Otezla fasted(B): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  EU-Otezla fed(C): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  US-Otezla fed(D): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  Japan-Otezla fasted(E): One Japan-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  The 5 treatments were separated by a washout period of at least 5 days.
- Japan-Otezla Fasted(E)/ EU-Otezla Fasted(A)/ US-Otezla Fed(D)/ US-Otezla Fasted(B)/ EU-Otezla Fed(C): Treatment sequence EADBC was applied with the following treatments:
  EU-Otezla fasted(A): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  US-Otezla fasted(B): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  EU-Otezla fed(C): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  US-Otezla fed(D): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
  Japan-Otezla fasted(E): One Japan-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
  The 5 treatments were separated by a washout period of at least 5 days.
Period: Overall Study
Arm/Group | EU-Otezla Fasted(A)/ Japan-Otezla Fasted(E)/ US-Otezla Fasted(B)/ US-Otezla Fed(D)/ EU-Otezla Fed(C) | US-Otezla Fasted(B)/ EU-Otezla Fasted(A)/ EU-Otezla Fed(C)/ Japan-Otezla Fasted(E)/ US-Otezla Fed(D) | EU-Otezla Fed(C)/US-Otezla Fasted(B)/US-Otezla Fed(D)/EU-Otezla Fasted(A)/ Japan-Otezla Fasted(E) | US-Otezla Fed(D)/ EU-Otezla Fed(C)/ Japan-Otezla Fasted(E)/ US-Otezla Fasted(B)/ EU-Otezla Fasted(A) | Japan-Otezla Fasted(E)/ US-Otezla Fed(D)/ EU-Otezla Fasted(A)/EU-Otezla Fed(C)/ US-Otezla Fasted(B) | EU-Otezla Fasted(A)/ US-Otezla Fasted(B)/ Japan-Otezla Fasted(E)/ EU-Otezla Fed(C)/ US-Otezla Fed(D) | US-Otezla Fasted(B)/ EU-Otezla Fed(C)/ EU-Otezla Fasted(A)/ US-Otezla Fed(D)/ Japan-Otezla Fasted(E) | EU-Otezla Fed(C)/ US-Otezla Fed(D)/ US-Otezla Fasted(B)/ Japan-Otezla Fasted(E)/ EU-Otezla Fasted(A) | US-Otezla Fed(D)/ Japan-Otezla Fasted(E)/ EU-Otezla Fed(C)/ EU-Otezla Fasted(A)/ US-Otezla Fasted(B) | Japan-Otezla Fasted(E)/ EU-Otezla Fasted(A)/ US-Otezla Fed(D)/ US-Otezla Fasted(B)/ EU-Otezla Fed(C)
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set includes all subjects who were randomized and treated with at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | EU-Otezla Fasted(A)/ Japan-Otezla Fasted(E)/ US-Otezla Fasted(B)/ US-Otezla Fed(D)/ EU-Otezla Fed(C) | US-Otezla Fasted(B)/ EU-Otezla Fasted(A)/ EU-Otezla Fed(C)/ Japan-Otezla Fasted(E)/ US-Otezla Fed(D) | EU-Otezla Fed(C)/US-Otezla Fasted(B)/US-Otezla Fed(D)/EU-Otezla Fasted(A)/ Japan-Otezla Fasted(E) | US-Otezla Fed(D)/ EU-Otezla Fed(C)/ Japan-Otezla Fasted(E)/ US-Otezla Fasted(B)/ EU-Otezla Fasted(A) | Japan-Otezla Fasted(E)/ US-Otezla Fed(D)/ EU-Otezla Fasted(A)/EU-Otezla Fed(C)/ US-Otezla Fasted(B) | EU-Otezla Fasted(A)/ US-Otezla Fasted(B)/ Japan-Otezla Fasted(E)/ EU-Otezla Fed(C)/ US-Otezla Fed(D) | US-Otezla Fasted(B)/ EU-Otezla Fed(C)/ EU-Otezla Fasted(A)/ US-Otezla Fed(D)/ Japan-Otezla Fasted(E) | EU-Otezla Fed(C)/ US-Otezla Fed(D)/ US-Otezla Fasted(B)/ Japan-Otezla Fasted(E)/ EU-Otezla Fasted(A) | US-Otezla Fed(D)/ Japan-Otezla Fasted(E)/ EU-Otezla Fed(C)/ EU-Otezla Fasted(A)/ US-Otezla Fasted(B) | Japan-Otezla Fasted(E)/ EU-Otezla Fasted(A)/ US-Otezla Fed(D)/ US-Otezla Fasted(B)/ EU-Otezla Fed(C) | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.5 (13.4) | 43.5 (13.4) | 40.5 (7.8) | 30.5 (14.8) | 38.0 (18.4) | 39.5 (3.5) | 25.0 (2.8) | 48.5 (7.8) | 30.5 (4.9) | 43.5 (2.1) | 38.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 7
  Male | 0 | 2 | 2 | 1 | 1 | 2 | 2 | 1 | 2 | 0 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Apremilast in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: The area under the concentration-time curve of apremilast in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported.
Time Frame: 1 hour (h) before and 30 minutes (min), 1h, 1h30min, 2h, 2h30min, 3h, 3h30min, 4h, 5h, 6h, 8h, 11h, 15h, 24h, 36h, 48h after study drug administration.
Population: Pharmacokinetic (PK) set: This set includes all subjects in the treated set (TS) who provide at least one PK endpoint that was defined as primary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * nanogram / milliliter (h*ng/mL)
Groups:
- EU-Otezla Fasted (A; Tfasted): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
- US-Otezla Fasted (B; R1fasted): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
- EU-Otezla Fed (C; Tfed): One EU-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
- US-Otezla Fed (D; R1fed): One US-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fed state (after a high-fat, high-calorie meal).
- Japan-Otezla Fasted (E; R2fasted): One Japan-sourced Otezla® film-coated tablet of 30 milligrams (mg) apremilast was administered orally with 240 milliliter (mL) water as a single dose in the fasted state (after an overnight fasting period of at least 10 hours (h)).
Arm/Group | EU-Otezla Fasted (A; Tfasted) | US-Otezla Fasted (B; R1fasted) | EU-Otezla Fed (C; Tfed) | US-Otezla Fed (D; R1fed) | Japan-Otezla Fasted (E; R2fasted)
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
hour * nanogram / milliliter (h*ng/mL) | 2390 (39.5) | 2430 (35.5) | 2580 (35.6) | 2580 (39.6) | 2350 (36.9)

2. Primary Outcome: Area Under the Concentration-time Curve of Apremilast in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: The area under the concentration-time curve of apremilast in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * nanogram / milliliter (h*ng/mL)
Arm/Group | EU-Otezla Fasted (A; Tfasted) | US-Otezla Fasted (B; R1fasted) | EU-Otezla Fed (C; Tfed) | US-Otezla Fed (D; R1fed) | Japan-Otezla Fasted (E; R2fasted)
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
hour * nanogram / milliliter (h*ng/mL) | 2420 (39.3) | 2460 (35.4) | 2600 (35.6) | 2600 (39.6) | 2370 (36.9)

3. Primary Outcome: Maximum Measured Concentration of Apremilast in Plasma (Cmax)
Description: The maximum measured concentration of apremilast in plasma (Cmax) is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram / milliliter (ng/mL)
Arm/Group | EU-Otezla Fasted (A; Tfasted) | US-Otezla Fasted (B; R1fasted) | EU-Otezla Fed (C; Tfed) | US-Otezla Fed (D; R1fed) | Japan-Otezla Fasted (E; R2fasted)
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
nanogram / milliliter (ng/mL) | 298 (36.1) | 301 (35.6) | 303 (27.8) | 271 (39.0) | 299 (33.0)

ADVERSE EVENTS:
Time Frame: For serious and non-serious adverse events: From drug administration until end of residual effect period of 4 days, up to 5 days for each treatment group. For all-cause mortality: From drug administration until end of follow-up period, up to 11 days for each treatment group.
Description: Treated set (TS): The treated set includes all subjects who were randomized and treated with at least one dose of study drug.
Arm/Group | EU-Otezla Fasted (A; Tfasted) | US-Otezla Fasted (B; R1fasted) | EU-Otezla Fed (C; Tfed) | US-Otezla Fed (D; R1fed) | Japan-Otezla Fasted (E; R2fasted)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 1/20 | 3/20 | 5/20 | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EU-Otezla Fasted (A; Tfasted) (N=20) | US-Otezla Fasted (B; R1fasted) (N=20) | EU-Otezla Fed (C; Tfed) (N=20) | US-Otezla Fed (D; R1fed) (N=20) | Japan-Otezla Fasted (E; R2fasted) (N=20)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 2 | 3

LIMITATIONS AND CAVEATS:
This trial was prematurely discontinued due to sponsor decision. The planned recruitment amount was not reached. The planned statistical analyses of the pharmacokinetic parameters were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT04811573/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT04811573/SAP_001.pdf